CLINICAL TRIAL: NCT06393244
Title: Effectiveness of a Theory-based Home-based Multi-component Exercise Training Among Older Adults With Type 2 Diabetes Mellitus: Study Protocol of a Sequential Mixed-methods Study
Brief Title: A Theory-based Home-based Multi-component Exercise Training Among Older Adults With Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cheng Li (Other)
Responsible Party: Sponsor-Investigator, Cheng Li, Associate Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: L2023SYSU-HL-052
Record Dates: First submitted 2024-04-23; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus Type 2; Sarcopenia
Keywords: Type 2 diabetes mellitus; The risk of developing Sarcopenia; Multi-component exercise program; Interaction model of client health behavior
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sarcopenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Experimental): a theory-based home-based multi-component exercise training
  Interventions: Behavioral: a theory-based home-based multi-component exercise training
- the waiting list control group (No Intervention): the waiting list control

INTERVENTIONS:
Behavioral: a theory-based home-based multi-component exercise training — The participants in the intervention group will receive a 12-week theory-based home-based MCE program, which consists of three phases: exercise mobilization phase, exercise preparation phase (exercise instructions and exercise plan determination), and home-based autonomous exercise training. Structured guidelines have been developed for the intervention by the research team. This allowed interveners to deliver the intervention in a structured way with the same dosage.
  Arms: the intervention group

SUMMARY:
The goal of this clinical trial is to learn if a theory-based home-based multi-component exercise training works to prevent sarcopenia in older adults with type 2 diabetes mellitus. It will also learn about the safety of the theory-based home-based multi-component exercise training. The main questions it aims to answer are:

* Whether a 12-week theory-based home-based MCE program is effective in decreasing the risk of developing sarcopenia, as well as improving physical activity, glycaemic control, muscle mass, muscle strength, physical performance, cognitive function, depressive mood, and quality of life among the Chinese community-dwelling older patients with T2DM.
* What are the underlying mechanisms of the exercise intervention.

Researchers will compare the MCE program to a waiting list control group to see if the MCE program works to prevent sarcopenia.

Participants will:

· Take a MCE program or a waiting list for 6 months

DETAILED DESCRIPTION:
Background: Despite international consensus and guidelines recommend multi-component exercise for the older adults to improve their physical function and quality of life. There is a paucity of research exploring the effectiveness and the mechanisms of multi-component exercise in older patients with type 2 diabetes mellitus.

Aim: To evaluate the effectiveness of a 12-week theory-based home-based multi-component exercise program for Chinese community-dwelling older adults with type 2 diabetes mellitus, and to clarify the underlying mechanisms of the exercise intervention in this population.

Design: This study adopted a sequential mixed-methods design comprising a prospective, two-arm, assessor-blinded randomised controlled trial and a descriptive qualitative study.

Methods: A total of 96 eligible patients will be recruited from a community health service center in Guangzhou, China. And they will be randomly assigned to the intervention group or the waiting list control group with block randomization at a 1:1 ratio after baseline measurement. Participants in the intervention group will receive a 12-week theory-based home-based multi-component exercise program. The primary outcomes are the risk of sarcopenia and physical activity. Secondary outcomes include glycaemic control (measured by FBG and HbA1c), muscle mass, muscle strength, physical performance, cognitive function, depressive mood, quality of life. Data will be collected at baseline (T0), post-intervention (T1), 3 months after the intervention (T2). Intervention effects will be analyzed using the generalized estimating equation model on the basis of the intention-to-treat principle. For the qualitative study, individual semi-structured interviews will be conducted with some participants based on maximum variation principle in the intervention group. Content analysis methods will be used to analyze the qualitative data to explore the underlying mechanisms of the intervention.

Discussion: This study is expected to provide an effective and practical intervention to prevent or control sarcopenia among Chinese community-dwelling older adults with type 2 diabetes mellitus. The results of this study will demonstrate the effectiveness and potential mechanisms of multicomponent exercise, contributing to the existing evidence in this filed.

Impact: This study will provide useful evidence for health professionals to provide health care and early intervention for older patients with T2DM to prevent or control sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* are community-dwelling older adults aged 60 years or above and have been diagnosed with T2DM;
* are able to communicate in Chinese;
* have a smartphone to receive intervention materials and messages;
* provide written informed consent for voluntary participation in this study.

Exclusion Criteria:

* meet the AWGS 2019 diagnostic criteria for sarcopenia;
* are currently participating in any other exercise intervention program or within the last 6 months;
* have any contraindication to exercise training according to the American College of Sports Medicine (ACSM) or are medically prohibited from participating in exercise;
* have a history of cognitive disorders or psychopathy, as identified in their medical records;
* severe visual or hearing problems,

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
the risk of developing sarcopenia | baseline, 3 months, 6 months
  The change of the scores of Strength, Assistance with Walking, Rise from a Chair, Climb Stairs and Falls (SARC-F) or Assistance with Walking, Rise from a Chair, Climb Stairs and Falls, Calf Circumference (SARC-CalF) or calf circumference (CC) among older adults with type 2 diabetes mellitus during the intervention period and follow-up period. The SARC-F consists of 5 items, which total scores ≥4 points can be judged as patients with high risk of developing sarcopenia. The total scores of SARC-CalF range from 0 to 20, with total scores ≥11 points indicating patients with high risk of developing sarcopenia. AWGS 2019 recommends CC <34cm for males and CC <33cm for females to indicate a high risk of developing sarcopenia among Asian populations.
the level of physical activity | baseline, 3 months, 6 months
  The change of the scores of physical activity scale for the elderly (PASE) among older adults with type 2 diabetes mellitus during the intervention period and follow-up period. This scale comprises 10 items across three dimensions: leisure, housework, and occupational physical activity. The total scores range from 0 to 500, with higher total scores indicating higher physical activity among the older adults.

SECONDARY OUTCOMES:
Fasting blood glucose (FBG) | baseline, 3 months, 6 months
  The change of fasting blood glucose among older adults with type 2 diabetes mellitus during the intervention period and follow-up period. The blood samples of participants will be collected by community health service center nurses early in the morning after fasting overnight (at least 8h), for FBG. All determinations will be performed in the same laboratory at the community health service center. FBG will be measured using enzymatic colorimetric assay.
muscle mass, | baseline, 3 months, 6 months
  The change of the scores of muscle mass among older adults with type 2 diabetes mellitus during the intervention period and follow-up period. Bioelectrical impedance analyzer (BIA) is widely used to measure muscle mass in older adults in the community because it is affordable, widely available and portable. A multi-frequency BIA, InBody 120 will be used to estimate body composition including appendicular skeletal muscle mass (ASM). As muscle mass is related to body size, muscle mass will be assessed using the appendicular skeletal muscle mass index (ASMI) (kg/m2), which is height-squared adjusted ASMM.
muscle strength | baseline, 3 months, 6 months
  The change of handgrip strength among older adults with type 2 diabetes mellitus during the intervention period and follow-up period. A digital handgrip strength dynamo-meter will be used to measure handgrip strength in participants. The participants will be instructed to assume a standing position with their hands naturally placed at the side of the body. The dominant and non-dominant hands are then measured twice, with the maximum value recorded.
physical performance | baseline, 3 months, 6 months
  The change of the scores of short physical performance battery (SPPB) among older adults with type 2 diabetes mellitus during the intervention period and follow-up period. The SPPB is a comprehensive tool for testing physical performance, including three parts: balance test, 4-meter walking speed test and 5-time sitting test. The total scores range from 0 to 12, with higher total scores indicating higher physical function among older adults.
cognitive function | baseline, 3 months, 6 months
  The change of the scores of montreal cognitive assessment (MoCA) among older adults with type 2 diabetes mellitus during the intervention period and follow-up period. The MoCA contains 12 items across cognitive tasks for a range of domains, including episodic memory, visuospatial ability, executive function, attention, language and orientation to obtain an overview of one's cognitive function. The total scores range from 0 to 30, with higher total scores indicating better cognitive function.
depressive mood | baseline, 3 months, 6 months
  The change of the scores of 15-item geriatric depression scale (GDS-15) among older adults with type 2 diabetes mellitus during the intervention period and follow-up period. The GDS-15 scale comprises 15 dichotomous questions that describe the primary symptoms of depression, including reduced satisfaction with life, decreased interest in activities, a sense of emptiness in life, loss of hope for the future, decreased energy, and more. The total scores range from 0 to 15, with higher scores indicating more severe depressive symptoms.
EQ-5D-5L | baseline, 3 months, 6 months
  The change of the scores of EuroQol five-dimensional five-level questionnaire (EQ-5D-5L) among older adults with type 2 diabetes mellitus during the intervention period and follow-up period. The EQ-5D-5L comprises five dimensions: mobility (MO), self-care (SC), usual activities (UA), pain/discomfort (PD), and anxiety/depression (AD), each dimension is described at five levels (corresponding roughly to no, slight, moderated, severe, and extreme problems). The total scores range from 0 to 100, with lower total scores indicating better quality of life.
Hemoglobin A1c (HbA1c) | baseline, 3 months, 6 months
  The change of hemoglobin A1c (HbA1c) among older adults with type 2 diabetes mellitus during the intervention period and follow-up period. The blood samples of participants will be collected by community health service center nurses early in the morning after fasting overnight (at least 8h), for HbA1c. All determinations will be performed in the same laboratory at the community health service center. HbA1c will be measured using high-performance liquid chromatography (AKRAY HA 8180V, Menarini Diagnostics).

CONTACTS AND LOCATIONS:
Locations (1):
- Yuexiu District Baiyun Street community health service center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The non-identified IPD will be shared after outcomes have been published.
Supporting Information: SAP
Time Frame: After the publication of the study
Access Criteria: Researchers should contact the PI for approval of the study protocol.